CLINICAL TRIAL: NCT07047222
Title: Behavioral Change Communication Intervention in Menstrual Disorder Management Among Female University Students in Bangladesh
Brief Title: Improving Menstrual Health Through BCC Among Bangladeshi University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahjalal University of Science and Technology (Other)
Responsible Party: Principal Investigator, G.M. Rabiul Islam, principal investigator (PI) of the study, Shahjalal University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AST/002/258
Record Dates: First submitted 2025-06-08; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Dysmenorrhea; Premenstrual Syndrome-PMS; Menstrual Irregularity
Keywords: Menstrual Health; Menstrual disorders; Behavior Change Communication; Lifestyle Intervention; Female University Students; BCC Module; Dietary Diversity; Physical Activity; Bangladesh; Propensity Score Matching (PSM)
MeSH Terms: conditions — Dysmenorrhea; Premenstrual Syndrome; Menstruation Disturbances; Motor Activity

STUDY DESIGN:
Intervention Model Description: The BCC module aimed to enhance awareness and promote effective management of menstrual disorders through structured guidance on lifestyle and behavioral changes. It included three sessions: the first covered menstrual disorders and their associated risk factors, the second focused on dietary habits, and the third addressed physical activity (including yoga) and other lifestyle factors. Sessions were conducted from May 20 to June 30, 2023, at PSTU, BU, and KU in Bangladesh by two trained female educators. Informed consent was obtained from interested participants. Session dates were approved by university authorities and included presentations, yoga demonstrations, pamphlet distribution, quizzes, and gifts. Participants were followed up every two months from July 15, 2023, to January 15, 2024, to support behavior change. A quasi-experimental post-evaluation (Feb-Mar 2024) used dormitory records and propensity score matching to compare outcomes with a control group.
Masking Description: This was a quasi-experimental study with non-random recruitment conducted through campus outreach and voluntary registration. Interested students who wished to participate in BCC module were invited to register by providing their name, contact number, room number, residence name, and university. To form the control group, an equal number of students from the same residences who did not participate in the BCC sessions were identified and listed. Since participation in the intervention was voluntary and based on personal interest, random sampling was neither feasible nor aligned with the study objectives. Therefore, participants were selected using purposeful, non-random sampling based on their characteristics and willingness to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Female university students who voluntarily registered for the structured BCC module formed the intervention group. The module comprised three interactive sessions that combined educational presentations, yoga demonstrations, distribution of informative pamphlets, quiz-based learning, and the provision of small rewards to encourage active engagement. To support lasting behavior change and address any ongoing challenges, follow-up sessions were conducted every two months.
  Interventions: Behavioral: Behavioral change communication (BCC) module
- Control group (No Intervention): The Control group consisted of female students from the same universities who did not receive any educational session of BCC module or follow-up during the intervention period. They were selected using student dormitory records and matched to the intervention group through propensity score matching to ensure comparability. As they did not receive any form of intervention, this group served as the matched comparison group for evaluating the effectiveness of the BCC module on menstrual health outcomes.

INTERVENTIONS:
Behavioral: Behavioral change communication (BCC) module — The behavior change communication (BCC) module was designed to enhance awareness and promote effective management of menstrual disorders through structured lifestyle and behavioral guidance. It consisted of three 1-hour sessions: (1) education on menstrual disorders and related risk factors; (2) healthy dietary practices; and (3) physical activity (including yoga) and other lifestyle improvements. Sessions were held from May 20 to June 30, 2023, at three public universities in Bangladesh and were delivered by trained female educators. All session dates were approved by university authorities. Activities included interactive presentations, yoga demonstrations, pamphlet distribution, quizzes, and gift giveaways. To reinforce and support behavior change, follow-up visits were conducted every two months from July 15, 2023, to January 15, 2024.
  Other Names: BCC module
  Arms: Intervention group

SUMMARY:
This study evaluated the effectiveness of a Behavior Change Communication (BCC) intervention in improving menstrual health among female university students in Bangladesh. The intervention focused on three outcomes: dysmenorrhea, premenstrual syndrome (PMS), and menstrual irregularity (MI), promoting a non-pharmacological, sustainable approach through behavioral and lifestyle changes.

Three structured educational sessions on menstrual health, healthy diet, and physical activity were delivered by trained female educators between May 20 and June 30, 2023, at Patuakhali Science and Technology University, Barishal University, and Khulna University. Participation was voluntary. Reinforcement follow-ups were conducted every two months for six months.

A quasi-experimental design was employed. Post-intervention data were collected from February to March 2024. Based on sample size calculations assuming a 30% reduction in disorder prevalence, 498 students (249 per group) were initially enrolled. After exclusions, 234 intervention and 238 control participants were analyzed for dysmenorrhea; 228 per group for PMS and MI. Propensity score matching (1:1, caliper 0.01, no replacement) yielded 98 matched participants per group for final analysis.

Eligible participants were female students aged ≥19 years, residing in university dormitories. Data collection used validated Bengali-language, interviewer-administered questionnaires, based on relevant literature and menstrual health IEC materials. Trained female enumerators ensured data quality and participant comfort.

Primary outcomes were: (1) Dysmenorrhea, measured by the Andersch and Milsom score (dichotomized Yes/No); (2) PMS, assessed using the Premenstrual Symptoms Screening Tool, with no/mild PMS and moderate to severe PMS/PMDD as the outcome; (3) MI, defined as self-reported menstrual cycles <21 or >35 days. The treatment variable was BCC exposure (Yes/No).

Covariates included physical activity, BMI, dietary diversity (DDS ≥5), food cravings, breakfast skipping, sleep duration, caffeine use, bedtime, family history of menstrual disorders, age at menarche, marital status, residence, and parental education and occupation.

Baseline differences were assessed using descriptive statistics, chi-square, and t-tests. Conditional logistic regression estimated intervention effects on matched data. Sensitivity analyses (ATE, ATT, balance diagnostics, Bayesian logistic regression) supported the robustness of results.

DETAILED DESCRIPTION:
This study aimed to assess the effectiveness of a structured Behavior Change Communication (BCC) intervention in improving menstrual health among female university students in Bangladesh. Specifically, it targeted three key menstrual health outcomes: dysmenorrhea, premenstrual syndrome (PMS), and menstrual irregularity (MI). The overarching goal was to promote a sustainable, non-pharmacological strategy for managing common menstrual disorders by fostering positive lifestyle and behavioral changes-such as healthier eating habits, increased physical activity, and greater awareness about menstrual health.

The study employed a quasi-experimental design involved two groups: an intervention group that received BCC module and a control group that did not. Participants were female undergraduate students at three public universities in Bangladesh i.e. Patuakhali Science and Technology University (PSTU), Barishal University (BU), and Khulna University (KU). Ethical approval was obtained from the Shahjalal University of Science and Technology Research Ethics Board (Ref. No. AST/002/258), and all participants provided written informed consent.

The BCC intervention comprised three interactive educational sessions delivered between May 20 and June 30, 2023, by trained female facilitators. The first session addressed menstrual disorders and associated risk factors, the second focused on healthy dietary practices, and the third emphasized physical activity (including yoga) and other relevant lifestyle modifications. To enhance retention and adherence, follow-up visits were conducted bi-monthly for six months after the intervention to reinforce key messages and address participant questions or barriers to behavior change. Post-intervention data collection was carried out between February and March 2024.

Participants were eligible if they were female students aged 19 years or older, residing full-time in university dormitories, and not currently taking hormonal treatments or diagnosed with chronic illnesses affecting menstruation. Recruitment occurred through record book of student dormitories at each university and student networks. Informed written consent was obtained prior to participation.

Data were collected through interviewer-administered questionnaires, adapted and validated in Bengali for cultural relevance and comprehension. Instruments were based on existing literature and government-endorsed information, education, and communication (IEC) materials on menstrual health. All interviews were conducted by trained female enumerators to ensure a comfortable and respectful environment for participants.

The sample size was calculated to detect a 30% reduction in the prevalence of menstrual disorders, with 80% statistical power and a 95% confidence interval, accounting for an anticipated dropout rate. Initially, 498 participants were recruited-249 each in the intervention and control groups. After excluding individuals with missing follow-up data or incomplete attendance, 234 participants in the intervention group and 238 in the control group were included in the analysis for dysmenorrhea. For PMS and MI outcomes, 228 participants per group had valid data.To control for potential confounding, 1:1 propensity score matching (PSM) was conducted using nearest-neighbor matching with a caliper of 0.01 and without replacement. Matching was based on baseline characteristics to ensure statistical equivalence between groups. After matching, a balanced analytical sample of 196 participants (98 in each group) was retained for all outcome analyses.

Among all the primary outcomes, dysmenorrhea was assessed using the Andersch and Milsom four-point scale and dichotomized as no pain (Grade 0) vs. any pain (Grades 1 - 3). PMS was evaluated by the premenstrual symptoms screening tool (PSST) and recoded into a binary variable: No/Mild PMS (code = 0) and Moderate to Severe PMS or premenstrual dysphoric disorder (PMDD) (code = 1). Additionally, Menstrual irregularity was determined based on self-reported cycle length and coded as irregular (1) if <21 or >35 days, and not irregular (0) if within the 21-35 day range.

The primary exposure variable was participation in the BCC intervention, coded as yes (intervention group) or no (control group).

The covariates included physical activity, obesity, dietary habits, lifestyle factors, and socio-demographic characteristics. Physical activity was classified according to WHO guidelines as: (i) sedentary: light-intensity activities; (ii) active: moderate-intensity activities for 150-300 minutes per week; and (iii) athlete: vigorous-intensity activities for 75-150 minutes per week. Obesity was assessed using body mass index (BMI, kg/m²) and categorized according to WHO Asian-specific cut-offs: (i) underweight (<18.5), (ii) normal weight (18.5-22.9), (iii) overweight (23.0-27.5), and (iv) obese (>27.5). Dietary information was evaluated through 24-hour dietary recall using FAO's Minimum Dietary Diversity for Women (MDD-W) scoring system, with scores ≥5 indicating adequate diversity was collected using a five-day 24-hour recall method, and dietary diversity score (DDS) was calculated following FAO guidelines. Lifestyle-related covariates included food cravings for high-fat or sweet foods, skipping breakfast, sleep duration, bedtime and caffeine intake. Socio-demographic variables included family history of menstrual disorders, age at menarche, marital status, and participants' residence as well as parental educational and occupational status.

Data analysis was performed using Stata 17. The following steps were undertaken:

1. Descriptive statistics summarized baseline demographic and behavioral characteristics. Chi-square (χ²) tests were used for categorical variables, and independent-sample t-tests for continuous variables.
2. Propensity score matching (PSM) was conducted using logistic regression to estimate the probability of receiving the intervention, based on the identified covariates. Nearest-neighbor matching (1:1) with a caliper width of 0.01 (no replacement) was applied. Balance between groups post-matching was assessed using standardized mean differences (SMD), with values <10% indicating adequate balance.
3. Primary analyses of intervention effects were conducted using conditional logistic regression on the matched sample to estimate odds ratios (ORs) and 95% confidence intervals (CIs) for each outcome.
4. To confirm the robustness of the findings, bivariate and multivariate logistic regression analyses were also performed on the unmatched sample, adjusting for covariates.
5. Sensitivity analyses were carried out to assess the stability of the results, including: covariate balance diagnostics (before and after matching); estimation of Average Treatment Effect (ATE) and Average Treatment Effect on the Treated (ATT); Bayesian logistic regression, including log Bayes factor interpretation, to evaluate model fit and strength of evidence for intervention effects. However, All statistical tests were two-sided, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Female university students aged 19 to 25 years, based on self-reported age, verified through enrollment records. The young adult female of this age range was selected to capture reproductive-aged participants most likely to experience menstrual disorders.
* Currently enrolled as full-time undergraduate students at one of the following selected public universities in Bangladesh: Patuakhali Science and Technology University (PSTU), Barisal University (BU), or Khulna University (KU). These institutions were selected based on logistical feasibility and representativeness of the target population.
* Willing and able to provide written informed consent after being fully informed of the study's purpose, procedures, potential risks, and benefits, and their rights as participants. Informed consent was obtained in accordance with ethical guidelines of SUST Research Ethics Board (SREB).
* Available and committed to participating in all phases of the study, including all three intervention sessions (BCC module), bimonthly follow-up over a six-month period (July 2023 to January 2024) and in evaluation of the intervention's effectiveness.
* Have regular access to a mobile phone, email, or another reliable means of communication to receive reminders, updates, and follow-up contacts related to intervention sessions and data collection.
* Able to comprehend and respond to study instructions and questionnaires in either Bengali or English, ensuring accurate data collection and meaningful engagement in the intervention.
* Not currently pregnant or breastfeeding, as confirmed during initial screening, to ensure hormonal stability and comparability across participants.

Exclusion Criteria:

* Currently receiving treatment with hormonal contraceptives, hormone replacement therapy, or any other medication specifically prescribed to manage menstrual disorders (e.g., dysmenorrhea, premenstrual syndrome, or irregular menstrual cycle).
* History of major abdominal or gynecological surgery (e.g., hysterectomy, oophorectomy, or myomectomy) that may affect menstrual function or reproductive physiology.
* Clinical diagnosis of chronic gynecological conditions, including but not limited to polycystic ovary syndrome (PCOS), endometriosis, or uterine fibroids.
* Diagnosed with chronic endocrine disorders such as thyroid disease, adrenal disorders, or diabetes mellitus, which may affect menstrual health.
* Pregnant, planning to conceive, or currently breastfeeding at the time of enrollment.
* Participation in another clinical trial or intervention study related to reproductive health, dietary habit, or physical activity.
* Presence of any diagnosed psychiatric illness or cognitive impairment that could interfere with participation in educational sessions or accurate reporting of menstrual symptoms.
* Refusal or inability to provide informed consent or commit to the follow-up schedule.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 498 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Dysmenorrhea | Participants received three BCC sessions over approximately 6 weeks, followed by regular support to encourage behavior change for up to 6 months, with monitoring every two months. Final outcomes were assessed about 8 months after enrollment.
  Dysmenorrhea pain was evaluated using a four-point grading scale that assessed both the severity of pain and its interference with the daily activities: Grade 0 indicated no pain, Grade 1 mild pain, Grade 2 moderate pain, and Grade 3 severe pain. For analytical purposes, this scale was dichotomized into a binary variable, where "0" represented the absence of pain (Grade 0), and "1" indicated the presence of any level of pain (Grades 1 to 3: mild, moderate, or severe).
Prevalence of Premenstrual syndrome (PMS) | Each participant received three BCC sessions over 6 weeks, followed by behavior change support and follow-up for 6 months. The final outcome evaluation was performed approximately 8 months after enrollment.
  Premenstrual symptoms were assessed using premenstrual symptoms screening tool (PSST) and categorized into three groups: No/Mild PMS, Moderate to Severe PMS, and premenstrual dysphoric disorder (PMDD). For analysis, these were combined into a binary variable: 0 = No/Mild PMS and 1 = Moderate to Severe PMS or PMDD
Prevalence of Menstrual Irregularity (MI) | Each participant completed the BCC sessions over approximately 6 weeks and followed by 6 months of support to encourage behavior change. The outcomes were assessed about 8 months after enrollment.
  Menstrual cycle irregularity was assessed based on participants' self-reported cycle lengths. A cycle was considered irregular (coded 1 = Yes) if it was shorter than 21 days or longer than 35 days. Cycles within the 21-35 day range were classified as not irregular (coded 0 = No)

CONTACTS AND LOCATIONS:
Overall Officials: GM Rabiul Islam, PhD, Principal Investigator — Shahjalal University of Science and Technology Research
Locations (1):
- Patuakhali Science and technology University, Dumki, Patuakhali, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary findings published from this study will be made available to qualified academic or public health researchers upon reasonable request. Shared data will include demographic characteristics and post-intervention outcomes on menstrual health (e.g., dysmenorrhea, premenstrual symptoms, irregular menstrual cycle); socio-demographic variables (e.g., age at menarche, residence, marital status, parental education/occupation, family history of menstrual disorders); lifestyle factors (e.g., physical activity, BMI, dietary diversity, food cravings, caffeine intake, sleep, bedtime); and group assignment (intervention vs. control). Associated data dictionaries and coding manuals will be provided. The IPD will be fully de-identified in accordance with data protection standards to ensure participant confidentiality. The goal is to support reproducibility, meta-analyses, and further research on menstrual health interventions.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will become available 6 months after publication of this study results in a peer-reviewed journal and will remain accessible for a duration of 3 years. During this availability period, qualified researchers affiliated with academic, governmental, or non-profit public health institutions may request access to the dataset to verify findings, conduct secondary analyses, or contribute to meta-analyses focused on menstrual health outcomes (e.g., dysmenorrhea, PMS, irregular menstrual cycles) among young adult female populations.
Access Criteria: Qualified researchers may request access to the data for academic, non-commercial purposes. Requests must include a detailed research proposal and will be reviewed by the principal investigator and ethics committee. Access will be granted only if the proposal is methodologically sound, aligns with the original consent, and ensures participant confidentiality. Approved researchers must sign a data use agreement to protect participant privacy and comply with all ethical and legal data use requirements.

REFERENCES:
- [Background] Mitsuhashi R, Sawai A, Kiyohara K, Shiraki H, Nakata Y. Factors Associated with the Prevalence and Severity of Menstrual-Related Symptoms: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Dec 29;20(1):569. doi: 10.3390/ijerph20010569. PMID 36612891
- [Background] Hanley-Cook GT, Tung JYA, Sattamini IF, Marinda PA, Thong K, Zerfu D, Kolsteren PW, Tuazon MAG, Lachat CK. Minimum Dietary Diversity for Women of Reproductive Age (MDD-W) Data Collection: Validity of the List-Based and Open Recall Methods as Compared to Weighed Food Record. Nutrients. 2020 Jul 9;12(7):2039. doi: 10.3390/nu12072039. PMID 32659995
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Ansong E, Arhin SK, Cai Y, Xu X, Wu X. Menstrual characteristics, disorders and associated risk factors among female international students in Zhejiang Province, China: a cross-sectional survey. BMC Womens Health. 2019 Feb 18;19(1):35. doi: 10.1186/s12905-019-0730-5. PMID 30777053
- [Background] Steiner M, Macdougall M, Brown E. The premenstrual symptoms screening tool (PSST) for clinicians. Arch Womens Ment Health. 2003 Aug;6(3):203-9. doi: 10.1007/s00737-003-0018-4. PMID 12920618
- [Background] Andersch B, Milsom I. An epidemiologic study of young women with dysmenorrhea. Am J Obstet Gynecol. 1982 Nov 15;144(6):655-60. doi: 10.1016/0002-9378(82)90433-1. PMID 7137249
- [Background] Sen LC, Jahan I, Salekin N, Shourove JH, Rahman M, Uddin MJ, Zhang C, H Hamer D, Islam GMR. Food craving, vitamin A, and menstrual disorders: A comprehensive study on university female students. PLoS One. 2024 Sep 25;19(9):e0310995. doi: 10.1371/journal.pone.0310995. eCollection 2024. PMID 39321166
- [Background] Slap GB. Menstrual disorders in adolescence. Best Pract Res Clin Obstet Gynaecol. 2003 Feb;17(1):75-92. doi: 10.1053/ybeog.2002.0342. PMID 12758227
- [Background] Rupe ER, Rodean J, Hurley EA, Miller MK, Boncoeur MD, Masonbrink AR. Menstrual health among adolescents and young adults in rural Haiti. Reprod Health. 2022 Dec 20;19(1):227. doi: 10.1186/s12978-022-01533-4. PMID 36539795

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT07047222/Prot_SAP_ICF_000.pdf